CLINICAL TRIAL: NCT01601327
Title: Effects of Three Different Medications on Metabolic Parameters and Testicular Volume in Patients With Hypogonadotropic Hypogonadism-Last Three Years Experience
Brief Title: Effects of Medications in Patients With Hypogonadism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Aydogan Aydogdu, Principal Investigator, Gulhane School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 01052012
Record Dates: First submitted 2012-05-01; First posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Idiopathic Hypogonadotropic Hypogonadism
Keywords: hypogonadism; treatment; testis volume
MeSH Terms: conditions — Idiopathic Hypogonadotropic Hypogonadism; Hypogonadism | interventions — testosterone enanthate; Testosterone; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypogonadism, treatment (Other): 77 patients with idiopathic hypogonadotropic hypogonadism were treated with testosterone gel, testosterone enanthate or human chorionic gonadotropin
  Interventions: Drug: Testosterone enanthate (Sustanon 250 mg); Drug: Human chorionic gonadotropin (hCG) (Pregnyl 5000 IU); Drug: Testosteron gel (Testojel 50 mg)
- Control group (No Intervention): 42 healthy controls
  Interventions: Drug: Testosterone enanthate (Sustanon 250 mg)

INTERVENTIONS:
Drug: Testosterone enanthate (Sustanon 250 mg) — Twenty-eight patients were treated with testosterone enanthate (TE),
Drug: Human chorionic gonadotropin (hCG) (Pregnyl 5000 IU) — twenty-five patients were treated with human chorionic gonadotropin (hCG)
  Arms: hypogonadism, treatment
Drug: Testosteron gel (Testojel 50 mg) — Twenty-four patients were treated with testosterone gel (TG).
  Arms: hypogonadism, treatment

SUMMARY:
The aim of the present study was to demonstrate the influences of three different treatment strategies on biochemical parameters and testicular volume (TV) in patients with idiopathic hypogonadotropic hypogonadism (IHH).

ELIGIBILITY:
Inclusion Criteria: hypogonadotropic hypogonadism

* decreased serum testosterone concentration below the normal range (serum T < 300ng/dL),
* FSH and LH levels within or below the normal range,
* absence of a pituitary or hypothalamic mass lesions on MRI, presence of gonadotropin response to repetitive doses of GnRH,
* normal smell test and normal karyotypes

Exclusion Criteria:

* previous androgen treatment,
* history of smoking,
* presence of bilateral anorchia,
* intellectual deficiency,
* diabetes mellitus,
* arterial hypertension or dyslipoproteinemia,
* medication of any kind and drug abuse. Because of possible confounding effects, patients with other hormone deficiencies were excluded.

Participants with iron, vitamin B12 or folate deficiency were also excluded.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2008-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Effects of testosterone enanthate and testosterone gel on BMI, haemoglobin, haematocrit, urea creatinine, triglyceride, total testosterone (TT) and HDL-cholesterol were measured. | 3 years
Effects of testosterone gel on BMI, haemoglobin, haematocrit, urea creatinine, triglyceride, total testosterone (TT) and HDL-cholesterol were measured. | 3 years
Effects of human chorionic gonadotrophin on BMI, haemoglobin, haematocrit, urea creatinine, triglyceride, total testosterone (TT) and HDL-cholesterol were measured. | 3 years

SECONDARY OUTCOMES:
Effect of testosterone enanthate on testis volumes | 3 years
Effect of testosterone gel on testis volumes | 3 years
Effect of human chorionic gonadotrophin on testis volumes | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Aydogan Aydogdu, MD, Principal Investigator — Gulhane School of Medicine, Department of Endocrinology and Metabolism
Locations (2):
- Turkey (Türkiye) (2):
  - Gulhane School of Medicine Dep. of Endocrine and Metabolism, Ankara
  - Gulhane School of Medicine Dep. of Endocrinology and Metabolism, Ankara